CLINICAL TRIAL: NCT06654921
Title: The Safety and Efficacy of Remote Ischemic Conditioning for the Treatment of Diabetic Kidney Disease: a Single-center Double-blinded Randomized Controlled Study
Brief Title: Remote Ischemic Conditioning for the Treatment of Diabetic Kidney Disease
Acronym: RIC-DKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIC-DKD
Record Dates: First submitted 2021-07-03; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Kidney Disease (DKD)
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIC group (Experimental): Subjects in the intervention group will receive remote ischemic conditioning and standard background medical treatment.
  Interventions: Device: Remote ischemic conditioning; Drug: Standard medication therapy
- Sham group (Sham Comparator): Subjects in the placebo group will receive sham remote ischemic conditioning and standard background medical treatment.
  Interventions: Device: Sham remote ischemic conditioning; Drug: Standard medication therapy

INTERVENTIONS:
Device: Remote ischemic conditioning — RIC is a non-invasive therapy that performed by an electric auto-control device with cuff placed on arm. RIC procedures consist of five cycles of 5-min inflation (200 mmHg) and 5-min deflation of cuff on bilateral arm. The procedure will be performed twice daily for consecutive 6 months after enrollment.
  Other Names: RIC
  Arms: RIC group
Device: Sham remote ischemic conditioning — Sham RIC will be performed by the same electric auto-control device with cuff placed on arm. Sham RIC procedures consist of five cycles of 5-min inflation (60 mmHg) and 5-min deflation of cuff on bilateral arm. The procedure will be performed twice daily for consecutive 6 months after enrollment.
  Other Names: Sham RIC
  Arms: Sham group
Drug: Standard medication therapy — Standard medication therapy will be performed according to the national and international guidelines.

SUMMARY:
Chronic kidney disease (CKD) is a growing epidemic affecting 10% of the population worldwide. Significantly, diabetic kidney disease (DKD) is the main cause of CKD and affects approximately 40% of patients with diabetes. Approximately 10% of patients with early-stage CKD and approximately half of patients with advanced-stage CKD suffer progression to renal failure and require dialysis or transplantation to survive. Moreover, DKD progresses particularly rapidly and has a poor prognosis, accounting for almost 50% of end-stage renal disease (ESRD) cases. Dialysis in particular is a burdensome therapy associated with poor patient outcomes and high societal and economic costs. Clinical studies using RIP have demonstrated protection against ischemic target renal damage in a variety of acute and chronic clinical settings . In the renal setting, RIP performed in dialysis patients is known to abrogate brain, heart and liver ischemia occurring during hemodialysis treatments. RIP may play a role in reducing the incidence of cardiac surgery-associated acute kidney injury. However, whether RIP can improve the renal function of patients with DKD is unclear and is worthy of further study.

Our overarching hypothesis is that RIP, performed in DKD patients, could delay progression to renal failure by abrogating progressive ischemic damage in the failing kidney. The present proposal is a pilot study addressing this hypothesis and is aimed at generating proof-of-concept and feasibility data on the benefits of RIP in patients with DKD.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a growing epidemic affecting 10% of the population worldwide. Significantly, diabetic kidney disease (DKD) is the main cause of CKD and affects approximately 40% of patients with diabetes. Approximately 10% of patients with early-stage CKD and approximately half of patients with advanced-stage CKD suffer progression to renal failure and require dialysis or transplantation to survive. Moreover, DKD progresses particularly rapidly and has a poor prognosis, accounting for almost 50% of end-stage renal disease (ESRD) cases. Dialysis in particular is a burdensome therapy associated with poor patient outcomes and high societal and economic costs. Strategies to prevent progression to renal failure focus on exquisite blood pressure control, renin-angiotensin-aldosterone system (RAAS) inhibition for proteinuria DKD, and glycemic control with the use of sodium-glucose cotransporter-2 (SGLT-2) inhibitors in patients with diabetes. Even so, despite the optimization of these parameters, many high-risk DKD patients will progress to renal failure. Recurrent ischemic damage to the failing and fibrotic kidney appears to be one of the final common pathways of progressive kidney damage in late-stage DKD, irrespective of the original cause of kidney disease. Specific strategies to alter this pathway in DKD have not yet been developed. In this context, it is crucial to seek novel pharmaceutical or nonpharmaceutical approaches to optimize the treatment of DKD.

With the progression of DKD, renal interstitial fibrosis intensifies, leading to severe ischemia and hypoxia of kidney cells and ultimately leading to ESRD. Therefore, effectively delaying the process of renal fibrosis can slow or even reverse the process of DKD. Hypoxia is characterized by an insufficient supply of oxygen to organs, and hypoxia-inducible factor (HIF) regulates gene transcription in hypoxia. Appropriate renal hypoxia can activate HIF-1α and suppress HIF-2α, improving the ability of the kidney to adapt to hypoxia, reducing transforming growth factor (TGF)-β pathway activity and further inhibiting fibrosis development. Therefore, increasing the expression of HIF-1 in renal tissue may be a new method to delay renal interstitial fibrosis and the progression of DKD to ESRD. Previous studies have provided evidence that HIF-1α participates in remote ischemic preconditioning (RIP). HIF-1α levels are significantly increased in the peripheral blood after RIP is implemented. Therefore, we speculated that RIP may have a therapeutic effect on DKD.

Ischemic conditioning occurs when a transient episode of ischemia reduces the effect of a subsequent larger ischemic insult. Similar levels of protection can be achieved by RIP. RIP is a noninvasive physical therapy that induces remote vital organs to adapt to ischemia through repeated, short-term ischemia-reperfusion training on nonvital organs such as limbs, thereby improving their tolerance to ischemic injury and enabling them to withstand subsequent fatal ischemic events. Clinical studies using RIP have demonstrated protection against ischemic target renal damage in a variety of acute and chronic clinical settings. In the renal setting, RIP performed in dialysis patients is known to abrogate brain, heart and liver ischemia occurring during hemodialysis treatments. RIP may play a role in reducing the incidence of cardiac surgery-associated acute kidney injury. However, whether RIP can improve the renal function of patients with DKD is unclear and is worthy of further study.

Our overarching hypothesis is that RIP, performed in DKD patients, could delay progression to renal failure by abrogating progressive ischemic damage in the failing kidney. The present proposal is a pilot study addressing this hypothesis and is aimed at generating proof-of-concept and feasibility data on the benefits of RIP in patients with DKD.

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 diabetes and receiving at least 1 antidiabetic medication
* CKD at stage G3 or G4 (eGFR = 15-60 mL/min/1.73 m2)
* UACR ≥ 300 mg/g or urinary albumin excretion rate (UAER) ≥ 300 mg/24 h
* Patients are cognitively and physically capable and willing to interact with the device and perform self-measurements
* Ability to withstand 5 full minutes of cuff inflation during prescreening

Exclusion Criteria:

* Patients with New York Heart Association Class III or IV congestive heart failure at enrollment
* Patients with severe illness with an expected lifespan of less than 6 months
* Patients with a recent history (< 6 months) of continuous renal replacement therapy, malignant tumor, myocardial infarction, acute coronary syndrome, stroke, seizure, thrombotic/thromboembolic event (e.g., deep vein thrombosis or pulmonary embolism), or a cerebrovascular accident
* Patients with known severe arterial disease of the extremities (ulcers, amputations, known symptomatic peripheral arterial disease)
* Patients at imminent risk of starting dialysis during the study period
* Patients residing in a long-term care facility
* Patients in another interventional trial that could influence the intervention or outcome of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The tolerability of RIC in patients with DKD | 0-6 months
  Patients who complete at least of twice a day up to 5 months of RIC treatment are considered to be tolerable of RIC.

SECONDARY OUTCOMES:
ΔSerum creatinine | 0-6 months
  Changes of serum creatinine before and after the intervention. Serum creatinine is one of biomarkers of CKD progression, which is tested in fasting serum.
ΔSerum Cystatin C | 0-6 months
  Changes of serum Cystatin C before and after the intervention. Serum Cystatin C is one of biomarkers of CKD progression, which is tested in fasting serum.
ΔHemoglobin | 0-6 months
  Changes of hemoglobin before and after the intervention. Hemoglobin is used to evaluate renal anemia in CKD patients.
ΔSerum KIM-1 | 0-6 months
  Changes of serum KIM-1 before and after the intervention. Serum kidney injury molecule-1 (KIM-1) is the biomarker of renal tubule injury.
ΔUrine microalbumin-creatinine ratio | 0-6 months
  Changes of urine microalbumin-creatinine ratio before and after the intervention. Urine microalbumin-creatinine ratio is the diagnostic as well as the disease progression biomarker of CKD.
ΔEstimated glomerular filtration rate | 0-6 months
  Changes of Estimated glomerular filtration rate before and after the intervention. Estimated glomerular filtration rate is calculated using the CKD-EPI equation by serum creatinine and Cystatin C.
ΔSerum VEGF | 0-6 months
  Changes of serum VEGF before and after the intervention. Serum vascular endothelial growth factor (VEGF) is related to the mechanism of RIC.
ΔSerum HIF-1 | 0-6 months
  Changes of serum HIF-1 before and after the intervention. Hypoxia inducible factor-1 (HIF-1) is related to the mechanism of RIC and CKD progression.
Δurine protein | 0-6 months
  Changes o furine protein before and after the intervention. Urine protein is related to the mechanism of RIC and CKD progression.
Incidence of major adverse cerebral and cardiac events | 0-6 months
  Myocardial infarction or stroke will be evaluated by professional investigators.
Incidence of Kidney failure | 0-6 months
  Clinical outcome; to observe the proportion of patients who requires dialysis or transplantation.
Incidence of all-cause death | 0-6 months
  Clinical outcome; to observe the proportion of all patients who died in each group.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bello AK, Levin A, Tonelli M, Okpechi IG, Feehally J, Harris D, Jindal K, Salako BL, Rateb A, Osman MA, Qarni B, Saad S, Lunney M, Wiebe N, Ye F, Johnson DW. Assessment of Global Kidney Health Care Status. JAMA. 2017 May 9;317(18):1864-1881. doi: 10.1001/jama.2017.4046. PMID 28430830
- [Background] Wakashima T, Tanaka T, Fukui K, Komoda Y, Shinozaki Y, Kobayashi H, Matsuo A, Nangaku M. JTZ-951, an HIF prolyl hydroxylase inhibitor, suppresses renal interstitial fibroblast transformation and expression of fibrosis-related factors. Am J Physiol Renal Physiol. 2020 Jan 1;318(1):F14-F24. doi: 10.1152/ajprenal.00323.2019. Epub 2019 Oct 21. PMID 31630548
- [Background] Wang Y, Meng R, Song H, Liu G, Hua Y, Cui D, Zheng L, Feng W, Liebeskind DS, Fisher M, Ji X. Remote Ischemic Conditioning May Improve Outcomes of Patients With Cerebral Small-Vessel Disease. Stroke. 2017 Nov;48(11):3064-3072. doi: 10.1161/STROKEAHA.117.017691. Epub 2017 Oct 17. PMID 29042490
- [Background] Ekeloef S, Homilius M, Stilling M, Ekeloef P, Koyuncu S, Munster AB, Meyhoff CS, Gundel O, Holst-Knudsen J, Mathiesen O, Gogenur I. The effect of remote ischaemic preconditioning on myocardial injury in emergency hip fracture surgery (PIXIE trial): phase II randomised clinical trial. BMJ. 2019 Dec 4;367:l6395. doi: 10.1136/bmj.l6395. PMID 31801725
- [Background] Zarbock A, Schmidt C, Van Aken H, Wempe C, Martens S, Zahn PK, Wolf B, Goebel U, Schwer CI, Rosenberger P, Haeberle H, Gorlich D, Kellum JA, Meersch M; RenalRIPC Investigators. Effect of remote ischemic preconditioning on kidney injury among high-risk patients undergoing cardiac surgery: a randomized clinical trial. JAMA. 2015 Jun 2;313(21):2133-41. doi: 10.1001/jama.2015.4189. PMID 26024502
- [Background] Li H, Satriano J, Thomas JL, Miyamoto S, Sharma K, Pastor-Soler NM, Hallows KR, Singh P. Interactions between HIF-1alpha and AMPK in the regulation of cellular hypoxia adaptation in chronic kidney disease. Am J Physiol Renal Physiol. 2015 Sep 1;309(5):F414-28. doi: 10.1152/ajprenal.00463.2014. Epub 2015 Jul 1. PMID 26136559
- [Derived] Wang L, Jia L, Huang S, Ren C, Yu Y, Wang Y, Zhao W, Ji X, Li S. Safety and efficacy of remote ischaemic preconditioning in diabetic kidney disease: a pilot randomised, parallel-arm, sham-controlled trial protocol. BMJ Open. 2025 Sep 3;15(9):e096851. doi: 10.1136/bmjopen-2024-096851. PMID 40903083